CLINICAL TRIAL: NCT05138081
Title: Comparative Effects of Proprioceptive Neuromuscular Facilitation Stretching and Stabilization Exercises of Upper Trapezius on Pain, Range of Motion and Functional Disability in Mobile Phone Users With Neck Pain
Brief Title: PNF Techniques Versus Stabilization Exercises of Trapezius Muscle PNF Techniques Verus Stabilization Exercises of Trapezius Muscle
Acronym: ROM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/862-1/2021
Record Dates: First submitted 2021-11-03; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: parallel assignment
Who Masked: Participant
Masking Description: single blinding
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF Stretching: Group A (Experimental): Routine physical therapy treatment
  Interventions: Other: PNF stretching
- Stabilization Exercises: Group B (Experimental): Routine physical therapy treatment
  Interventions: Other: Stabilization

INTERVENTIONS:
Other: PNF stretching — Neck flexion pattern The therapist slightly pulled the chin so that it was lifted and causing the neck to extend. Commands such as "pull your chin in" and "look at your left hip" were given to the patient. Resistance was given against left rotation, flexion and lateral flexion along with the traction to the patient's chin.Neck extension pattern The therapists lightly pulled the chin so that the neck was flexed; head was rotated and tilted to the left. Commands such as "lift your chin and then "lift your head to look above were given to the patient. Passive resistance was provided against right rotation, extension and lateral flexion.
  Arms: PNF Stretching: Group A
Other: Stabilization — Stabilization exercises are shoulder rolls, shrugging, chin tuck, scapular retraction, cervical extension. This was done for 15 repetition
  Arms: Stabilization Exercises: Group B

SUMMARY:
This project will compare the effects of Proprioceptive Neuromuscular Facilitation Stretching and Stabilization of Upper Trapezius on Pain, Range of Motion and Functional Disability in Mobile Phone User with mobile phone-induced Neck Pain. The population sample will be 50 divided randomly into two groups by concealed envelop method. Then I will collect data from the social security hospital Physiotherapy department, Lahore. Group A was given stretching exercises and Group B was given stabilization exercises (25 stretchings and 25stabilization). NDI and NPRS were used as an outcome measure to quantify the upper trapezius on pain, range of motion, and functional disability with non-specific neck pain.

DETAILED DESCRIPTION:
This project will compare the effects of Proprioceptive Neuromuscular Facilitation Stretching and Stabilization of Upper Trapezius on Pain, Range of Motion and Functional Disability in Mobile Phone User with mobile phone-induced Neck Pain. The population sample will be 50 divided randomly into two groups by concealed envelop method. Then I will collect data from the social security hospital Physiotherapy department, Lahore. Group A was given stretching exercises and Group B was given stabilization exercises (25 stretchings and 25stabilization). NDI and NPRS were used as an outcome measure to quantify the upper trapezius on pain, range of motion, and functional disability with non-specific neck pain. Single blinding of accessor was done at the time of recording of outcome measures pre and post-treatment Baseline was 4th week and 8th week. Eighty female participants and twenty male participants in each group. The duration was 9 months. The 18-30 years age range of both males and females were considered. There was not any statistically significant difference between the two groups as p > 0.05. But within-group changes show that there was a significant change in baseline, 4th week, and 8th-week readings for NDI, NPRS, and ROM with p < 0.05.

ELIGIBILITY:
Inclusion Criteria

* Male and female, age range 18-30years with non-specific neck pain.

  * Permanently mobile users spent more than 8 hours per day using their mobiles
  * Participants are willing to participate in the research.
  * Having constant or frequent neck pain of more than 4weeks duration.

Exclusion Criteria:

* Specific disorders of the cervical spine, such as disc prolapse, spinal stenosis, postoperative conditions in the neck and shoulder areas.

  * History of severe trauma, instability, spasmodic torticollis, migraine (frequency more than twice per month).
  * Peripheral nerve entrapment, fibromyalgia, hypermobility syndrome, shoulder diseases (tendonitis, bursitis, capsulitis).
  * Inflammatory rheumatic diseases, severe psychiatric illness, and other diseases that prevent physical loading, pregnancy, and other on-going therapies.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-28 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | baseline, 4th week, 8th week
  Pain will be measured by Numeric Pain rating scale. 000. NPRS is one of the ways to quantify pain and is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 no pain to 10 worst imaginable pain. It has been shown that a composite scoring system including best, worse, and current level of pain. Pain by definition is an unpleasant sensation and emotional experience that is related to tissue damage

SECONDARY OUTCOMES:
Functional Disability Index | baseline, 4th week, 8th week
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain.
  The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain 0affects a patient's daily life and to assess the self-rated disability of patients with neck pain.We currently know that the NDI consists of one factor - "physical disability" - although NDI scores correlate well with SF-36 mental component scores as well Functional disability has been defined as acquired difficulty in performing basic everyday tasks or more complex tasks needed for independent living. The Neck Disability Index (NDI) is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Ashraf, ms-msk, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Amoudi M, Ayed A. Effectiveness of stretching exercise program among nurses with neck pain: Palestinian perspective. Sci Prog. 2021 Jul-Sep;104(3):368504211038163. doi: 10.1177/00368504211038163. PMID 34459689
- [Background] Javdaneh N, Molayei F, Kamranifraz N. Effect of adding motor imagery training to neck stabilization exercises on pain, disability and kinesiophobia in patients with chronic neck pain. Complement Ther Clin Pract. 2021 Feb;42:101263. doi: 10.1016/j.ctcp.2020.101263. Epub 2020 Nov 19. PMID 33276225
- [Background] Kuo YL, Lee TH, Tsai YJ. Evaluation of a Cervical Stabilization Exercise Program for Pain, Disability, and Physical Impairments in University Violinists with Nonspecific Neck Pain. Int J Environ Res Public Health. 2020 Jul 28;17(15):5430. doi: 10.3390/ijerph17155430. PMID 32731521
- [Background] Jung SI, Lee NK, Kang KW, Kim K, Lee DY. The effect of smartphone usage time on posture and respiratory function. J Phys Ther Sci. 2016 Jan;28(1):186-9. doi: 10.1589/jpts.28.186. Epub 2016 Jan 30. PMID 26957754